CLINICAL TRIAL: NCT06786702
Title: A Prospective Analysis of the Effects of Round Ligament Preservation and Division in Laparoscopic Transabdominal Preperitoneal Inguinal Hernia Repair in Women.
Brief Title: The Importance of Preserving the Round Ligament in the Repair of Inguinal Hernias in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammet Mustafa Vural (Other Government)
Responsible Party: Sponsor-Investigator, Muhammet Mustafa Vural, assistant doctor, Başakşehir Çam & Sakura City Hospital
Organization: Başakşehir Çam & Sakura City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSH-GC-MMV-1
Record Dates: First submitted 2024-08-18; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Inguinal Hernia; Femoral Hernia; Obturator Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Hernia, Obturator

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective investigation focusing on women with inguinal hernias. Patients will be divided into two groups based on the management of the round ligament during laparoscopic TAPP (Trans Abdominal Pre-Peritoneal) hernia repair:
  Group 1: Patients in this group will have their round ligament preserved using different preservation techniques, specifically through a longitudinal incision technique in the peritoneum.
  Group 2: Patients in this group will have their round ligament cut close to the peritoneum using an energy device for sealing.
  Patients will be randomized into these groups, starting with the first patient assigned to Group 1. Each subsequent patient will be alternately assigned to the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Round Ligament Preservation) (Active Comparator): Patients will undergo laparoscopic TAPP surgery with the round ligament preserved. The preservation will be achieved using a longitudinal incision technique in the peritoneum.
  Interventions: Procedure: Laparoscopic TAPP (Trans Abdominal Pre-Peritoneal) hernia repair: Round Ligament Preservation
- Group 2 (Round Ligament Cutting) (Active Comparator): Patients will undergo laparoscopic TAPP surgery with the round ligament cut close to the peritoneum using an energy device.
  Interventions: Procedure: Laparoscopic TAPP (Trans Abdominal Pre-Peritoneal) hernia repair: Round Ligament Cutting

INTERVENTIONS:
Procedure: Laparoscopic TAPP (Trans Abdominal Pre-Peritoneal) hernia repair: Round Ligament Preservation — Group 1 (Round Ligament Preservation): Patients will undergo laparoscopic TAPP surgery with the round ligament preserved. The preservation will be achieved using a longitudinal incision technique in the peritoneum.
  Arms: Group 1 (Round Ligament Preservation)
Procedure: Laparoscopic TAPP (Trans Abdominal Pre-Peritoneal) hernia repair: Round Ligament Cutting — Group 2 (Round Ligament Cutting): Patients will undergo laparoscopic TAPP surgery with the round ligament cut close to the peritoneum using an energy device.
  Arms: Group 2 (Round Ligament Cutting)

SUMMARY:
The aim of this study is to evaluate the impact of preserving or not preserving the round ligament during laparoscopic Trans Abdominal Pre-Peritoneal (TAPP) hernia repair on postoperative outcomes in female patients. Specifically, the study will compare outcomes such as postoperative pain, seroma, hematoma, prolapsus of uterina , recurrence rates, and quality of life between patients whose round ligament was preserved versus those whose ligament was cut.

DETAILED DESCRIPTION:
Study Overview:

The aim of this study is to evaluate the impact of preserving or not preserving the round ligament during laparoscopic Trans Abdominal Pre-Peritoneal (TAPP) hernia repair on postoperative outcomes in female patients. Specifically, the study will compare outcomes such as postoperative pain, seroma, hematoma, prolapsus of uterina, recurrence rates, and quality of life between patients whose round ligament was preserved versus those whose ligament was cut.

Background:

In women, inguinal hernias are less common but can present as femoral, inguinal, or obturator hernias. Treatment usually involves surgical repair, which can be performed using open or laparoscopic techniques. Laparoscopic methods, especially TAPP and Total Extraperitoneal (TEP), are increasingly preferred due to their lower recurrence rates and other benefits compared to open surgery.

Advantages of Laparoscopic TAPP Surgery:

Small Incisions: Results in less risk of complications and cosmetic benefits. Bilateral Viewing: Allows visualization and treatment of both sides simultaneously.

Lower Infection Risk: Smaller incisions reduce the risk of infection. Faster Recovery: Less postoperative pain and quicker return to daily activities.

Reduced Recurrence: More effective in preventing recurrence, especially after an initial open surgery.

Round Ligament Considerations:

The round ligament connects the uterus to the labia majora and can be involved in the TAPP procedure. The debate centers on whether to preserve or cut the round ligament during surgery. Preservation can be technically challenging due to adhesions, but cutting the ligament might impact recurrence rates and patient outcomes negatively.

There is ongoing debate about whether to preserve or cut the round ligament during laparoscopic preperitoneal repair in female patients. Many surgeons express concerns that preserving the round ligament may increase the risk of hernia recurrence. A recent study encompassing 1,365 women who underwent various methods of inguinal hernia repair (open, laparoscopic, or robotic) found that in 868 cases (63.6%) , the round ligament was cut. This suggests that in practice, round ligament division is commonly performed during both open and laparoscopic procedures.

However, literature indicates that there are few studies with weak evidence suggesting that not preserving the round ligament may lead to issues such as pain, dyspareunia (pain during intercourse), organ prolapse, and decreased quality of life.

Study Objectives:

Compare Outcomes: Assess the effects of preserving versus cutting the round ligament on postoperative pain, hernia recurrence, and quality of life.

Prospective Analysis: Collect and analyze data prospectively to determine the optimal surgical approach.

Conclusion:

This study aims to provide insights into the optimal surgical technique for female inguinal hernia repair using TAPP, highlighting the importance of round ligament management and its impact on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For patients applying to the General Surgery Clinic of Basaksehir Cam Sakura City Hospital:
* Age Range: Female patients aged between 18 and 70 years.
* Type of Hernia: Patients with inguinal, direct or indirect, femoral, and obturator hernias.
* Surgical Indication: Patients indicated for TAPP (Transabdominal Preperitoneal) surgery.
* Consent: Patients who consent to participate in the study.
* General Anesthesia: Patients who are suitable for general anesthesia.
* Follow-up: Patients who attend follow-up appointments regularly.

Exclusion Criteria:

* Age: Female patients under 18 years old or over 70 years old.
* Surgical Technique: Patients who are operated on with techniques other than TAPP (e.g., TEP, conventional surgery).
* Hernia Type: Patients with strangulated or incarcerated hernias.
* Hernia Location: Patients with hernias outside the groin region.
* Surgical Site: Surgeries performed in different clinics.
* Gender: Male patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication | 1 years
  "Number of Participants with Postoperative Complications : Seroma (in centimeters) , Hematoma (in centimeters) , Loss of Sensation on Neurological Examination , Prolapse (in centimeters) Numbness (reported in anamnesis), Tingling (reported in anamnesis), Urinary Retention (reported in anamnesis), Dyspareunia (reported in anamnesis) . Measured at Day 1, Month 3, and Year 1"

SECONDARY OUTCOMES:
Duration of Operation (in minutes) | Per-operation
  Outcome Description:
  The total duration of the surgical operation, measured in minutes, recorded during the operation.
Blood Loss During Operation (in milliliters) | Per-operation
  Outcome Description:
  The amount of blood loss recorded during the operation, measured in milliliters.
Number of Tackers Used During Operation | Per-operation
  Outcome Description:
  The total number of tackers used during the operation.
Mesh Size Used in Operation (in square centimeters) | Per-operation
  Outcome Description:
  The size of the mesh used during the operation, measured in square centimeters.
Pain Score at the Hernia Side (Using EuraHS-QoL) | Measurements will be conducted on Day 1, at Month 3, and at Year 1
  Pain score assessed using the EuraHS-quality-of-life questionnaire, specific to the hernia side. The score reflects the level of pain experienced postoperatively.
Score for Activity Limitation Due to Pain or Discomfort (Using EuraHS-QoL) | Measurements will be conducted on Day 1, at Month 3, and at Year 1
  Activity limitation due to pain or discomfort in the hernia area, assessed using the EuraHS-quality-of-life questionnaire
Cosmetic Discomfort Score (Using EuraHS-QoL) | Measurements will be conducted on Day 1, at Month 3, and at Year 1
  Cosmetic discomfort related to the hernia area, assessed using the EuraHS-quality-of-life questionnaire. The score evaluates patient satisfaction with the cosmetic outcome

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet M. Vural, M.D, Principal Investigator — Basakşehir Çam Sakura Şehir Hastanesi
Locations (1):
- Başakşehir Çam Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renshaw S, Collins C, Gupta A, Poulose B, Haisley KR. Round Ligament Management in Female Patients Undergoing Inguinal Hernia Repair: Should We Divide or Preserve? J Am Coll Surg. 2022 Jun 1;234(6):1193-1200. doi: 10.1097/XCS.0000000000000207. Epub 2022 Apr 8. PMID 35703818